CLINICAL TRIAL: NCT01542814
Title: Acquisition of Mammography Images for Clinical Evaluation of FUJIFILM 3Dimensional Mammography
Brief Title: Collection of FUJIFILM's 3Dimensional Mammograms
Acronym: 3DM
Status: Completed | Type: Observational
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMSU2011-003A
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: Screening Mammogram; Diagnostic Mammogram; Benign; Malignant; BI-RADS Categories
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fujifilm 3Dimensional Mammography: Group of subjects being given Fujifilm 3D Mammography Imaging
  Interventions: Device: 2D FFDM
- 2D FFDM: Group of Subjects receiving FujiFilm or other FDA Approved 2D Mammography Imaging
  Interventions: Device: 3Dimensional Mammography

INTERVENTIONS:
Device: 3Dimensional Mammography — The FUJIFILM 3DM examination is a 4-view mammogram which includes CC and MLO views of each breast. For each view, a routine (0-degree) mammogram will be acquired followed immediately in the same compression by a second mammogram offset at 4 degrees.
  Other Names: FUJIFILM 3Dimensional Mammography
  Groups: 2D FFDM
Device: 2D FFDM — Standard of care screening mammogram.
  Groups: Fujifilm 3Dimensional Mammography

SUMMARY:
This image-acquisition study is designed to acquire the study image data and establish and document the clinical findings for each subject. The acquired data will be used to support FUJIFILM protocol FMSU2011-003B (Clinical Evaluation of FUJIFILM 3Dimensional Digital Mammography) and future regulatory submissions.

DETAILED DESCRIPTION:
This is an image acquisition reader study to observe differences between 3D FujiFilm Mammography and 2D approved Mammography

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Any ethnic or racial origin.
* Must come through the study via the screening or diagnostic pathway described above.
* Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.
* Meet none of the exclusion criteria.

Exclusion Criteria:

* • Presence of a breast implant.

  * Women with only a single breast; for example, post mastectomy patients.
  * Is pregnant or believes she may be pregnant.
  * A woman who has delivered and who has expressed the intention to breast-feed or is currently breast-feeding.
  * A woman who has significant existing breast trauma.
  * Have self-reported severe non-focal or bilateral breast pain affecting subject's ability to tolerate mammography examinations.
  * A woman who has had a mammogram performed for the purpose of therapy portal planning.
  * Inadequate technical quality mammography images, such as insufficient anatomical coverage or significant motion artifacts.
  * Cannot, for any known reason, undergo follow-up mammography examinations (where clinically indicated) at the participating institution.
  * Is an inmate (see US Code of Federal Regulations 45CFR46.306).

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects who are appearing for a routine screening examination or have been referred for further diagnostic evaluation after a screening examination (within 45 days) or have a 4-view mammogram (within 45 days) due to clinical concerns will be eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Acquire screening cases with and without breast cancer. | 18-months

CONTACTS AND LOCATIONS:
Overall Officials: Carl J. D'Orsi, MD, Principal Investigator — Emory University Healthcare
Locations (3):
- United States (3):
  - Scottsdale Medical Imaging, Limited (SMIL), Scottsdale, Arizona
  - Emory University Healthcare, Atlanta, Georgia
  - Elizabeth Wende Breast Care, LLC (EWBC), Rochester, New York